CLINICAL TRIAL: NCT05701046
Title: Anterior vs Posterior Surgery for Lumbar Isthmic Spondylolisthesis: Multicenter Prospective Cohort Study
Brief Title: Anterior vs Posterior Surgery for Lumbar Isthmic Spondylolisthesis
Status: Recruiting | Type: Observational
Sponsor: University of British Columbia (Other)
Responsible Party: Principal Investigator, Charlotte Dandurand, Spinal Neurosurgeon, University of British Columbia
Other Study IDs: H22-00699
Record Dates: First submitted 2023-01-03; First posted 2023-01-27 (Actual); Last update posted 2024-05-09 (Actual); Status verified 2024-05

CONDITIONS: Isthmic Spondylolisthesis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Anterior and oblique interbody fusion (ALIF, OLIF + Posterior fixation (open or MIS) or stand-alone)
  Interventions: Procedure: Interbody fusion surgery
- Posterior interbody fusion (TLIF or PLIF) (open or MIS)
  Interventions: Procedure: Interbody fusion surgery

INTERVENTIONS:
Procedure: Interbody fusion surgery — Interbody fusion surgery

SUMMARY:
Currently there is no consensus on the best surgical treatment of patients with symptomatic isthmic spondylolisthesis (IS). Clinical equipoise exists amongst experienced clinicians on the various surgical techniques available.

This study will involve multiple phases to answer specific research questions comparing anterior and posterior interbody fusion in patients with lumbar isthmic spondylolisthesis. The primary end point will be 1-year proportions of patients reaching minimal clinically important difference (MCID) in terms of leg pain measured by NRS leg. The secondary endpoints will be predetermined moderate to severe AEs, reoperations for nonunion, symptomatic adjacent segment disease, radiological alignment correction and correlation with HRQOL as well as economic analysis at 1, 2, 5 and 10 years.

ELIGIBILITY:
Inclusion Criteria:

* Male or female aged 18 years or older (or who have reached the age of majority in the participating province)
* Require surgical treatment for a diagnosis of single-level lumbar isthmic spondylolisthesis, any grade, in the lumbar and lumbosacral spine.
* Are able to communicate in English or French
* Anterior interbody fusion group will be defined as having had an anterior or oblique approach with a synthetic cage insertion, interbody bone graft without cage or plate-screw construct with or without posterior rod-screw construct
* Posterior interbody fusion group will have only posterior approach procedure.

Exclusion Criteria:

* Previous spinal surgery
* Specific pathology at level above and below:

  * Degenerative anterolisthesis
  * Pars defect above or below index level

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Adult patients with lumbar isthmic spondylolisthesis requiring surgical treatment
Sampling Method: Probability Sample
Enrollment: 489 (Estimated)
Dates: Start 2023-01-05 (Actual); Primary Completion 2028-02-15 (Estimated); Study Completion 2038-02-15 (Estimated)

PRIMARY OUTCOMES:
Proportions of patients reaching MCID for NRS leg at 1 year | at 1 year follow-up
  Proportions of patients reaching MCID for NRS leg (>=3)

SECONDARY OUTCOMES:
Proportion of patients with any predefined adverse events | 3 month follow-up data
Reoperation due to nonunion at index level or adjacent segment disease | 1 year- 2 year -5 year -10 year follow-up data
Change in radiological parameters | 1 year- 2 year -5 year -10 year follow-up data
  Level, Labelle classification, Degree of translation, SVA, Lumbar lordosis, segmental lordosis, sacral and spinopelvic parameters,
Correlation between improvement in radiological parameters and patient reported outcomes | 1 year- 2 year -5 year -10 year follow-up data
Change in Patient's reported outcome (PRO) : Numeric pain rating scale for back pain | 1 year- 2 year -5 year -10 year follow-up data
Change in Patient's reported outcome (PRO) : Oswestry disability index | 1 year- 2 year -5 year -10 year follow-up data
Change in Patient's reported outcome (PRO) : EuroQoL 5 dimension (EQ5D) | 1 year- 2 year -5 year -10 year follow-up data
Change in Patient's reported outcome (PRO) : 12 item short form survey (SF12) | 1 year- 2 year -5 year -10 year follow-up data
Change in Patient's reported outcome (PRO) : Patient Health Questionnaire Depression Scale (PHQ-8) | 1 year- 2 year -5 year -10 year follow-up data

CONTACTS AND LOCATIONS:
Locations (1):
- Vancouver General Hospital, Vancouver, British Columbia, Canada

IPD SHARING:
Plan to Share IPD: Undecided